CLINICAL TRIAL: NCT06471894
Title: Study on the Neural Circuit Mechanism of Regulating GABA by Gut Microbiota in Inflammatory Bowel Disease Combined With Depression
Brief Title: Neural Circuit Mechanism of Inflammatory Bowel Disease Combined With Depression
Acronym: NCMOIBDCWD
Status: Not yet recruiting | Type: Observational
Sponsor: LanZhou University (Other)
Responsible Party: Principal Investigator, Jun Wang, Principal Investigator, LanZhou University
Other Study IDs: 2024A-255
Record Dates: First submitted 2024-06-18; First posted 2024-06-24 (Actual); Last update posted 2024-06-25 (Actual); Status verified 2024-06

CONDITIONS: Inflammatory Bowel Diseases
MeSH Terms: conditions — Inflammatory Bowel Diseases | interventions — FMT protocol

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — Fecal collection
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- CD: Crohn's disease
  Interventions: Radiation: Magnetic resonance imaging scanning; Drug: FMT Protocol
- UC: ulcerative colitis
  Interventions: Radiation: Magnetic resonance imaging scanning; Drug: FMT Protocol
- HC: healthy controls
  Interventions: Radiation: Magnetic resonance imaging scanning

INTERVENTIONS:
Radiation: Magnetic resonance imaging scanning — Perform brain diffusion imaging, magnetic resonance spectroscopy, and functional magnetic resonance imaging scans on all individuals
Drug: FMT Protocol — Treatment of disease groups (UC and CD) using prepared fecal microbiota transplantation solution
  Groups: CD; UC

SUMMARY:
The goal of this observational study is to understand the effects of gut microbiota dysbiosis treatment in patients with inflammatory bowel disease (IBD) combined with depression. The main question it aims to answer is:

Does fecal microbiota transplantation (FMT) improve depression symptoms in IBD patients by altering GABA levels in the medial prefrontal cortex?

Participants already undergoing fecal microbiota transplantation (FMT) as part of their regular medical care for IBD and comorbid depression will undergo regular assessments of GABA levels, gut microbiota, and depression symptoms for the duration of the study.

DETAILED DESCRIPTION:
The high incidence of inflammatory bowel disease (IBD) combined with depression increases the risk of disease recurrence and treatment failure. Previous research by our team has found a positive correlation between decreased levels of the inhibitory neurotransmitter γ-aminobutyric acid (GABA) in the medial prefrontal cortex of IBD patients and the severity of depression. However, the underlying pathological mechanisms remain unknown. Prior studies have suggested that GABA regulates activity within neural circuits in the brain, and the levels of GABA in the brain are influenced by the gut microbiota. Based on this premise, our study aims to treat gut microbiota dysbiosis in IBD patients with comorbid depression using fecal microbiota transplantation (FMT). Our team will analyze the correlation between changes in GABA levels in the medial prefrontal cortex and gut microbiota using techniques such as metagenomics, metabolomics, and magnetic resonance spectroscopy imaging. Additionally, resting-state functional magnetic resonance imaging (fMRI) is used to perform dynamic causal modeling of the neural circuit in the brain to elucidate the regulatory mechanism of GABA level changes on these circuits. Finally, the investigators will validate the research findings using a dextran sulfate sodium (DSS)-induced colitis mouse model to explore the neurochemical mechanisms underlying IBD comorbid with depression. The results of this study will not only provide a deeper understanding of the regulatory role of changes in brain GABA levels on neural circuits but also offer a theoretical basis for the use of fecal microbiota transplantation in treating gut microbiota dysbiosis in IBD patients and prevent complications such as depression.

ELIGIBILITY:
Inclusion Criteria:

aged 18-65 years right-handed active disease (CDAI score ≥150, Mayo score >2).

Exclusion Criteria:

previous brain surgery those with severe and unstable physical diseases those with contraindications for MRI who cannot tolerate long-duration MRI examinations.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The inflammatory bowel disease (IBD) combined with depression have increased psychological stress. Individuals with IBD often face prolonged physical discomfort and treatment challenges, which can lead to increased emotional burden and susceptibility to depression. IBD is a chronic condition requiring long-term management and treatment. These ongoing lifestyle changes and medical burdens may contribute to feelings of sadness and depression. In summary, depression is common among individuals with inflammatory bowel disease. It is important to monitor the mental health of patients during treatment and provide proactive psychological support and intervention when needed.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2024-07-01 (Estimated); Primary Completion 2024-07-01 (Estimated); Study Completion 2027-12-01 (Estimated)

PRIMARY OUTCOMES:
Magnetic resonance spectroscopy | 1 week before and 1 week after FMT
  Changes in GABA content in the prefrontal lobe of the brain
Magnetic resonance spectroscopy | 1 week before and 1 week after FMT
  Changes in alpha diversity and differential abundance of gut microbiota

CONTACTS AND LOCATIONS:
Overall Officials: Jun Wang, Doctor, Study Chair — The Second Hospital & Clinical Medical School, Lanzhou University

IPD SHARING:
Plan to Share IPD: Yes
After the data collection is completed, the collected gut microbiota data will be shared
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Around December 31, 2026
Access Criteria: Email the corresponding author with reasonable reasons for inquiry